CLINICAL TRIAL: NCT06617767
Title: The Effect of Reiki on Subjective Well-being, Happiness, and Some Metabolic Variables in Patients With Type-II Diabetes: Single-blind Randomized Controlled Trial
Brief Title: The Effect of Reiki in Patients With Type-II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Ulviye Özcan Yüce, Assistant Professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/5/2
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Reiki; well-Being; happiness; metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Participant
Masking Description: Participants were told that there were intervention and control groups in the study, but it was not explained which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki (Experimental): The Reiki group received 20 minutes of remote Reiki once a day for 4 consecutive days
  Interventions: Other: Reiki
- Control (No Intervention): No intervention was applied to the control group

INTERVENTIONS:
Other: Reiki — The Reiki group received distant Reiki application to their energy centers for 20 minutes, once a day, for 4 consecutive days, by researchers with Reiki Stage II training under the guidance of a researcher with the Usui Reiki Master & Teacher degree.
  Arms: Reiki

SUMMARY:
Aim: To evaluate the effects of Reiki on subjective well-being, happiness, and some metabolic variables in patients with Type-II diabetes.

DETAILED DESCRIPTION:
This study, designed as a randomized controlled trial with a pretest-posttest design, was conducted between September 2022 and August 2023 at the Internal Medicine clinic of Kanuni Sultan Süleyman Training and Research Hospital, Istanbul Provincial Health Directorate. The participants were voluntary individuals who had been diagnosed with Type-II Diabetes Mellitus at least 6 months prior, had a BMI ≥ 25kg/m² (overweight or obese), HbA1c ≥ 6.5%, were following a diabetes-specific diet or using oral antidiabetics, and were neither Reiki practitioners nor instructors. Randomization was used to assign participants to either the Reiki group or the control group. During the pretest, participants were asked to complete the Personal Information Form, the Subjective Well-Being Scale (SWS), and the OXFORD Happiness Scale (OHS). Pre-intervention fasting and postprandial blood glucose levels, HbA1c percentage, body mass index, LDL-HDL/total cholesterol, triglyceride levels, and blood pressure measurements were obtained from the patients' records and documented.The Reiki group received 20 minutes of remote Reiki once a day for 4 consecutive days, while no intervention was applied to the control group. The Subjective Well-Being Scale and OXFORD Happiness Scale were reapplied to both groups at the first and second months following the intervention, and the metabolic values, along with these scales, were measured again in the third month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type-II Diabetes Mellitus at least 6 months prior
* Had a BMI ≥ 25kg/m² (overweight or obese)
* HbA1c ≥ 6.5%

Exclusion Criteria:

* Being diagnosed with another disease and needing treatment during the data collection process
* Being a Reiki practitioner or instructor
* Using insulin for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Subjective Well-Being | 3 months
  The Subjective Well-Being Scale is a measurement tool developed to determine the subjective experiences and vitality levels of individuals in terms of feeling lively, energetic and alert, and is based on individuals providing information about themselves. The seven-item, 7-point Likert-type scale is ranked from 1 (Does not apply to me at all) to 7 (Completely applies to me), and participants are asked to determine the extent to which they agree with the statement in each item. The scores of all items in the scale can be added to obtain the individual's total subjective vitality score. The range of scores on the scale varies between 7 and 49. High scores on the scale indicate that the individual has a high level of subjective vitality.It is expected that the scores that the participants receive from this scale will increase in the final measurement.
Happiness | 3 months
  OXFORD Happiness scale is a 29-item, 6-point Likert-type scale (1-I completely disagree, 6-I completely agree) developed to measure happiness. A high score obtained from the scale indicates an increase in the level of happiness. The scale score range varies between 29-174. It is expected that the scores that the participants receive from this scale will increase in the final measurement.

SECONDARY OUTCOMES:
HbA1c (%) | 3 months
  HbA1c, is the main biomarker used to assess long-term glycaemic control in individuals with diabetes.In the final test, this value was targeted to be below the level recorded in the pre test in Reiki gruop.
Fasting blood glucose level (mg/dL) | 3 months
  Fasting blood glucose level is the level of glucose in the blood measured after at least 8 hours of overnight fasting.In the final test, this value was targeted to be below the level recorded in the pre test.
Postprandial blood glucose levels (mg/dl) | 3 months
  Postprandial blood sugar is the blood sugar level measured 2 hours after food intake (first bite). It should not be over 140 mg/dl.In the final test, this value was targeted to be below the level recorded in the first test.
Body mass index (kg/m2) | 3 months
  The study initially included individuals who were overweight or obese (BMI ≥ 25kg/m²). The aim was to reduce the body mass index of the participants in the Reiki group, measured in the post-test.
LDL-kolesterol (mg/dL) | 3 months
  The highest LDL (low density lipoprotein) level in the post-test measurements of individuals in the Reiki group was targeted to be 130 mg/dL.
HDL-kolesterol (mg/dL) | 3 months
  The lowest HDL (high density lipoprotein) level in the post-test measurements of individuals in the Reiki group was targeted to be 40 mg/dL for women and 50 mg/dL for men.
Total kolesterol (mg/dL) | 3 months
  The highest total kolesterol level in the post-test measurements of individuals in the Reiki group was targeted to be 200 mg/dL.
Triglyceride levels (mg/dL) | 3 months
  The highest triglyceride level in the post-test measurements of individuals in the Reiki group was targeted to be 150 mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- Yüce, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No